CLINICAL TRIAL: NCT05384639
Title: Simultaneous Dual-Task Cycling Exercise Training on Cognitive Function for the Elderly
Brief Title: Dual-task Cycling System on Cognitive Function for the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Innovation and Technology Commission, Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020.319
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual-task Group (Experimental)
  Interventions: Device: Dual-task Group
- Cycling Group (Active Comparator)
  Interventions: Device: Cycling Group
- Cognitive Group (Active Comparator)
  Interventions: Device: Cognitive Group

INTERVENTIONS:
Device: Dual-task Group — Participant will cycle and perform cognitive training simultaneously.
  Arms: Dual-task Group
Device: Cycling Group — Participant will cycle only.
  Arms: Cycling Group
Device: Cognitive Group — Participant will perform cognitive training only.
  Arms: Cognitive Group

SUMMARY:
This project aims to develop a new dual-task stationary cycling system that can monitor and provide feedback on the aerobic exercise intensity, while administrating appropriate cognitive trainings targeting various cognitive sub domains through a screen in front of the user.

The proposed system is designed to train the brain with cognitive tasks and the body with aerobic exercises at the same time. The difficulties of the cognitive tasks are controlled by the users' previous performances on these tasks so that they wouldn't be too easy nor too difficult. Similarly, the intensity of the aerobic exercise will be monitored through an optical encoder for the cycling cadence, two power meters for the force output on the two pedals, as well as a heart rate monitor for the users' physiological response. Constant feedback is being provided to the users so that they will exercise at the correct intensity to provide the greater cardiovascular and cognitive benefits.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MCI or cutoff at 2 < n < 16 th percentile MoCA score according to the level of education and age
* Sufficient cognitive ability to follow simple instructions
* Able to understand content and purpose of the study
* Conscious and in stable physical condition

Exclusion Criteria:

* Any additional medical or psychological condition that would affect their ability to comply with the study protocol, e.g., a significant orthopaedic or chronic pain condition; or
* Severe hip, knee or ankle contracture that would preclude the passive range of motion of the leg
* Uncontrolled Cardiac issues

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
The Montreal Cognitive Assessment, Hong Kong Version (HK-MoCA) | Within one month after the last training session

SECONDARY OUTCOMES:
Trail Making Test | Within one month after the last training session
6 Minutes Walk Test | Within one month after the last training session
5 times Sit to Stand | Within one month after the last training session
10 meters walk Test | Within one month after the last training session
Graded Heart-rate Assessment | Within one month after the last training session

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, The Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No